CLINICAL TRIAL: NCT03350074
Title: Influence of Hepatitis B Virus (HBV) Envelope Glycoprotein Characteristics on HBsAg Clearance on Anti-HBV Treatment by Nucleos(t)Ide Analogues
Brief Title: HBV Envelope Proteins Variability on HBs Antigen Clearance Under Nucleos(t)Ide Analogue Therapy
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: DC 2013-1801
Record Dates: First submitted 2017-09-29; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-09

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B virus; PreS/S variability; Anti-HBV treatment
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA VHB VIRUS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hepatitis B virus (HBV) infection remains difficult to eradicate with about 240 million people living with HBV chronic infection. HBsAg clearance, correlated with a good clinical prognosis, is difficult to achieve even with antiviral treatments (3-14 %). HBV envelope proteins are essential for entry into hepatocyte and are targeted by the immune system. Molecular characteristics of HBV envelope proteins may favour better viral fitness at the entry step into hepatocytes and/or HBV escape from host immunity. Here we investigated whether variability of HBV envelope proteins can contribute to the differential responses to anti-HBV treatment in patients with HBsAg clearance or persistence.

DETAILED DESCRIPTION:
Our study is a retrospective study of patients with chronic hepatitis B virus, selected exclusively at the University Hospital Center of Nancy in the Department of Hepato-Gastroenterology (HGE). the patient inclusion criteria were as follows: Adult patients with chronic hepatitis B, treated with nucleos(t)ide analogues, mono-infected with HBV (without co-infection with HCV, HIV and HDV). For each patient included, biological, clinical and therapeutic data were collected retrospectively. Patients with loss of viral load on treatment were included in this study. Among them, patients showed either a clearance of HBsAg on treatment ("responders") or the control patients showed a persistence of HBsAg on treatment ("non-responders", control patients).

ELIGIBILITY:
Inclusion Criteria:

* adults
* patients with chronic hepatitis B
* treated with nucleos(t)ide analogues
* mono-infected with HBV (without co-infection with HCV, HIV and HDV)

Exclusion Criteria:

* minor
* pregnant women
* patients with VHC or VHD

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Our study is a retrospective study of patients with chronic hepatitis B virus, selected exclusively at the University Hospital Center of Nancy in the Department of Hepato-Gastroenterology (HGE). the patient inclusion criteria were as follows: Adult patients with chronic hepatitis B, treated with nucleos(t)ide analogues, mono-infected with HBV (without co-infection with HCV, HIV and HDV). For each patient included, biological, clinical and therapeutic data were collected retrospectively. Patients with loss of viral load on treatment were included in this study. Among them, patients showed either a clearance of HBsAg on treatment ("responders") or the control patients showed a persistence of HBsAg on treatment ("non-responders", control patients).
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Clearance of Hepatitis B surface antigen (HBsAg) | May 2016 (manuscript Velay et al., 2016)
  Subgroup of patients infected by HBV genotype D

SECONDARY OUTCOMES:
Clearance of Hepatitis B surface antigen (HBsAg) | September 2017 (manuscript Eschlimann et al., 2017)
  Subgroup of patients infected by HBV genotype A